CLINICAL TRIAL: NCT02300246
Title: Clinical, Histological and Micro-computed Tomographic Evaluation of Neoformed Tissue in Post-extraction Sockets Covered With Platelet-rich Fibrin (PRF) Membrane: a Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Eliane dos Santos Porto Barboza (Unknown); Diogo Luz (Unknown); Denise Mandarino (Unknown)
Responsible Party: Principal Investigator, Vittorio Moraschini Filho, PhD, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UFederalFluminense
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Alveolar Socket Preservation
Keywords: alveolar socket preservation; tooth extraction; platelet concentrates; growth factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group (Experimental): Alveolar socket post-extraction covered with PRF
  Interventions: Procedure: Platelet-Rich Fibrin
- Control Group (No Intervention): Only clot (spontaneous healing)

INTERVENTIONS:
Procedure: Platelet-Rich Fibrin — Alveolar socket preservation with Platelet-Rich Plasma
  Arms: Test Group

SUMMARY:
The platelet-rich fibrin (PRF), belongs to a new generation of plasma concentrate with biomechanical processing simplified and without the need for handling blood biochemistry. Some studies have shown the potential of PRF in release growth factors assisting and accelerating the regeneration of soft tissues, however with contradictory results regarding the hard tissues. The aim of this study will be to evaluate through clinical analyzes, histomorphometric and micro-computed tomographic images, the dimensional changes, the quantity and the quality of the tissues formed socket after extractions that receive membranes of PRF. 15 sockets (test group) will receive a membrane of PRF after extraction and the other 15 (control group) received no biomaterial (spontaneous healing).

DETAILED DESCRIPTION:
1. Development methodology This study will be a randomized controlled and will be conducted according to the principles outlined in the Declaration of Helsinki regarding experiments on human beings. This work was submitted to the Ethics Committee, with the approval number: CAAE: 21317113.4.0000.5243. To ensure the quality of this randomized study, guidelines RCT-CONSORT checklist will be followed.
2. Selection of volunteers / sample The sample will consist of 30 human alveolar socket. Selected volunteers must agree to participate in the study signed an informed consent form and being willing to follow the guidelines and proposed timelines. The volunteers will be treated at the Dental Clinical Research Center of the Fluminense Federal University. The 30 teeth involved in this study should provide an indication of tooth extraction without treatment possibilities, determined by clinical and radiological examination.
3. Pre-Surgical Treatment Dental and medical case histories will be conducted on all volunteers. Initially, volunteers will be selected and diagnosed by clinical examination and periapical radiographic or cone beam tomographic to assess the need for tooth extraction. All volunteers will undergo basic periodontal therapy and oral hygiene instructions. Volunteers who have a risk factor for bacterial endocarditis will be medicated with Amoxicillin 2g single dose one hour before the procedure, and for those allergic to penicillin, will be prescribed 600g single dose of clindamycin one hour before procedure, as recommended by the American College of Cardiology. Laboratory tests, including blood pressure measurement, complete blood count, lipid profile, coagulation profile and complete fasting glucose will be required for all volunteers.
4. Surgical Procedures Plaster study models are made by molding with alginate in all volunteers, to enable construction of the measuring guides (templates) in acrylic. Also intraoral photographs will be held. Volunteers will undergo local anesthesia (2% with epinephrine Mepvacaína - 1: 100.00) for extraction of teeth. In all cases, the extractions will be performed in a minimally traumatic manner and without lifting flap with the aim of preservation tissues. Incisions intra-sulculares the free surfaces (buccal / lingual) and proximal (mesial / distal) will be performed with a scalpel blade 15C aiming the disruption of the periodontal fibers. The dislocation of the tooth will be conducted with a forceps, with subsequent removal of the tooth socket. After extraction, a rigorous inspection and curettage of the socket for the removal of granulation tissue will be held, followed by irrigation with sterile saline.

   Performed after extraction, will start to make themselves venous blood of volunteers himself for a qualified professional with the goal of achieving the PRF membrane. For this, will be collected with a sterile without anti-coagulant about 10 ml of blood from the median cubital vein (arm) syringe. It will be led immediately into a test tube and centrifuge for which will be calibrated to 2700 rpm for 12 minutes. After processing, three phases are arranged within a test tube. The fibrin clot is obtained between the layers of acellular layer of plasma and red blood cells. The same tube is carefully collected and manipulated to form a membrane which is sutured with 5.0 absorbable synthetic yarn (Vycril - Johnson & Johnson). The sutures are removed seven days after the procedure.

   The remaining fifteen sockets (control group) are not filled with any biomaterial (only clot). Volunteers will be instructed to rinse their mouths twice daily for 15 days with chlorhexidine gluconate 0.12%.

   Queries review will be conducted in the first week for suture removal and the subsequent second and fifth weeks.
5. Clinical Evaluation Prior to the extraction of both groups, the bands of keratinized gingiva buccal and lingual measures are the muco-gingival line to the gingival margin, with support from the UNC-15 periodontal probe, positioned on a template (stent ) acrylic resin. Furthermore, measurements of the gingival margin of the template, track keratinized gingiva and the measurement from the edge of the template edge bony ridge will be held in the regions mesial, buccal and distal of the buccal and lingual surfaces. For the evaluation of the thickness of the tissues, a surgical caliper located at 5mm from the gingival margin is used. The data collected will be immediately recorded by an assistant. Clinical evaluations will be performed prior to extraction (T1) and 120 days (T2).
6. Histomorphometric analysis At T2, an implant will be installed in the socket region. The surgical bone obtained during the discharge procedure for implant placement through a trephine measuring about 3mm in diameter, will be collected. It will be stored in buffered formaldehyde, decalcified in EDTA, dehydrated in ethanol and embedded in paraffin. Serial sections including the central portion of the bone cylinder will be prepared parallel to the long axis, with the standard microtome in 5mm. The sections are stained with hematoxylin and eosin. The analysis of the new tissue formed is evaluated in Leitz microscope equipped with image capture system. Morphometric measurements are evaluated to determine the proportion occupied by mineralized bone (lamellar bone, immature bone), osteoid tissue (connective tissue matrix rich in collagen and partially mineralized), bone marrow (adipocytes and vascular structures), fibrous tissue and tissue residual (tissue elements unidentified artifacts of preparation).
7. Micro-computed tomographics Representative non-decalcified samples will be scanned at a resolution of 18 x 18 x 18 voxels μc3 using a micro-Pxs5-928EA cone beam CT. The GEHC MicroView Plus ® Analysis software (GE Healthcare), will be used to create three-dimensional reconstructions (3D) bone tissue from the scan. The tissue to be analyzed is represented by all or fragments of tissue biopsy samples. The value scale in grayscale will be used in each biopsy by a single calibrated examiner and anonymous. The value of the average grayscale will be calculated and used as the representative to evaluate bone volume (BV) and the mineral content of the tissue value. The tissue mineral density will also be calculated.
8. Statistical analysis The results express the mean ± 95% CI. Mann-Whitney tests will be conducted. Will be considered as significant differences when P < 0.05. Nominal data will be evaluated by chi-square test. Alternatively, in case of no associates (extreme) values, the Fisher exact test will be used. Continuous variables are expressed as mean and standard deviation and analyzed for normal distribution using the Shapiro-Wilk test. The Student t or Mann-Whitney tests will be applied for normal and non-normal distribution, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Healthy patients with indication for dental extraction
* Teeth adjacent to the extraction site
* Patients willing to cooperate with the study and who have signed the informed consent form.

Exclusion Criteria:

* Patients showing periapical or periodontal infection
* Patients with severe systemic diseases
* Patients on medications such as chemotherapy, anticoagulants, corticosteroids, biphosphonates and drugs imunossupressivas
* Patients who have chronic diseases decompensated (e.g. hypertension, diabetes, rheumatic diseases, renal, and hepatic)
* Patients with bone diseases, metabolic (osteomalacia, hypocalcemia and hypercalcemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Dimensional changes of the alveolar crest. | 120 days
  Clinical examination, histological and micro-computed tomography analyses will be conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Vittorio Moraschini, Niterói, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Farina R, Bressan E, Taut A, Cucchi A, Trombelli L. Plasma rich in growth factors in human extraction sockets: a radiographic and histomorphometric study on early bone deposition. Clin Oral Implants Res. 2013 Dec;24(12):1360-8. doi: 10.1111/clr.12033. Epub 2012 Sep 24. PMID 22998461
- [Background] Suttapreyasri S, Leepong N. Influence of platelet-rich fibrin on alveolar ridge preservation. J Craniofac Surg. 2013 Jul;24(4):1088-94. doi: 10.1097/SCS.0b013e31828b6dc3. PMID 23851746
- [Background] Alissa R, Esposito M, Horner K, Oliver R. The influence of platelet-rich plasma on the healing of extraction sockets: an explorative randomised clinical trial. Eur J Oral Implantol. 2010 Summer;3(2):121-34. PMID 20623037
- [Result] Hauser F, Gaydarov N, Badoud I, Vazquez L, Bernard JP, Ammann P. Clinical and histological evaluation of postextraction platelet-rich fibrin socket filling: a prospective randomized controlled study. Implant Dent. 2013 Jun;22(3):295-303. doi: 10.1097/ID.0b013e3182906eb3. PMID 23644909